CLINICAL TRIAL: NCT05770232
Title: In Order to Explore the Risk Factors of VTE After Acute Thoracic Trauma, we Collected the Diagnosis and Treatment Information of 5774 Patients With Thoracic Trauma From 33 Hospitals in China, Retrospectively Analyzed the Risk Factors of VTE in Patients With Thoracic Trauma, and Established a Risk Prediction Model.
Brief Title: Retrospectively Analyze the Risk Factors of VTE in 5774 Patients With Thoracic Trauma From 33 Hospitals in China, and Established a Risk Prediction Model
Acronym: MCTTVTE
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Weigang Zhao, Attending Physician, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: multi-center thorax VTE
Record Dates: First submitted 2023-03-04; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Thorax Injuries; Embolism Vein; Embolism, Pulmonary; Rib Fractures
Keywords: venous thrombus embolism; Thorax Injuries; risk factors; prediction model
MeSH Terms: conditions — Thoracic Injuries; Pulmonary Embolism; Rib Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospectively analyze the risk factors of VTE in 5774 patients with thoracic trauma from 33 hospitals in China, and established a risk prediction model

DETAILED DESCRIPTION:
In order to explore the risk factors of VTE after acute thoracic trauma, we collected the diagnosis and treatment information of 5774 patients with thoracic trauma from 33 hospitals in China, retrospectively analyzed the risk factors of VTE in patients with thoracic trauma, and established a risk prediction model.

ELIGIBILITY:
Inclusion Criteria:

* admitted within three days of the chest trauma, VTE has not yet occurred, AIS score of thoracic injury was greater than or equal to 3, AIS score of other combined injuries was less than or equal to 2.

Exclusion Criteria:

* received preventive physical or chemical anticoagulation before admission, VTE occurred before admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-80 years of age who were admitted within 3 days of chest trauma, did not have VTE prior to admission and were not receiving prophylactic anticoagulation. The chest trauma AIS score of QI patients with multiple injuries was greater than or equal to 3, and the chest trauma score of other combined injuries was less than or equal to 2.
Sampling Method: Probability Sample
Enrollment: 5774 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
VTE | Peri-treatment period
  venous thrombus embolism, including pulmonary embolism and deep vein thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China